CLINICAL TRIAL: NCT06318767
Title: Predictive Value of Systolic Rise Time of the Plantar Arch on the Risk of Major Adverse Limb Events (MALE) and Major Adverse Cardiovascular Events (MACE) in Peripheral Artery Disease (PAD) at Critical Ischaemia Stage
Acronym: TAMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2023_843_0141
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Major Adverse Limb Events; Major Adverse Cardiovascular Events; Peripheral Artery Disease; Critical Limb Ischemia; Hemodynamic Measure
Keywords: major adverse limb events; major adverse cardiovascular events; peripheral artery disease; critical limb ischemia; hemodynamic measure
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hemodynamic measure of the Systolic Time Rise — The hemodynamic measure of the Systolic Time Rise will be added in the routine doppler echography, planned in preoperative, postoperative and at 6 months of following up. This measure is taken on the foot, with ultrasound probe.

SUMMARY:
Peripheral artery disease (PAD), vascular disease of atheromatous origin, is a frequent pathology, with a steady and significant increase in prevalence over the last decades. It has various symptoms ranging from mild arterial claudication to critical limb ischemia. The critical ischaemia stage in PAD is defined by rest pain or trophic disorders and is a special situation because of the number of cardiovascular deaths at 1 year (25%), 60% at 5 years and acute ischaemic recurrence at 1 year (25%).

It is a medico-surgical pathology. A haemodynamic marker is needed to monitor patients, as it is predictive of limb progression, cardiovascular events and mortality. The Systolic Rise Time (SRT) of the plantar footpad is a recently described haemodynamic measurement of proven value in the diagnosis of PAD. The aim of this study is to show the prognostic value of the Systolic Rise Time on Major Adverse Limb Events (MALE).

ELIGIBILITY:
Inclusion Criteria:

* patients at least 18 years old,
* willing and able to provide written informed consent,
* with documented atherosclerosis critical limb ischemia (pain rest and/or ulcer and gangrene manifestations)
* with hemodynamic measures (ankle pressure less than 50mmHg and/or TBI less than 30mmHg and/or TcPO2 less than 30 mmHg),
* followed or send to CHU Amiens Picardie, and eligible to chirurgical revascularization.

Exclusion Criteria:

* with non atherosclerosis arteriopathy,
* ineligible to the gold standard treatment such as the chirurgical revascularization,
* with life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
occurrence of limb ischemia | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No